CLINICAL TRIAL: NCT06342921
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II/III Study of the Safety and Efficacy of ADC189 Tablets in the Treatment of Influenza A Virus Infection/Influenza B Virus Infection in Adolescents and Adults
Brief Title: ADC189 Tablets on Influenza A Virus Infection/Influenza B Virus Infection
Acronym: ADC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiaxing AnDiCon Biotech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADC189-2022-01
Record Dates: First submitted 2024-03-12; First posted 2024-04-02 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-03

CONDITIONS: Safety Issues; Effect of Drug

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 15 mg (Experimental): 15 mg of ADC189 tablets Once during the whole study.
  Interventions: Drug: 15 mg ADC189
- 45 mg (Experimental): 45 mg of ADC189 tablets Once during the whole study.
  Interventions: Drug: 45 mg ADC189
- Placebo (Placebo Comparator): Once during the whole study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 15 mg ADC189 — Use only once during the whole study.
  Arms: 15 mg
Drug: 45 mg ADC189 — Use only once during the whole study.
  Arms: 45 mg
Drug: Placebo — Use only once during the whole study.
  Arms: Placebo

SUMMARY:
The goal of this Phase II/III study is to investigate the safty and efficacy of ADC189 tablets in adolescents and adults with influenza A virus infection/influenza B virus infection.

The main aim to answer:

* Phase II study is to evaluate the efficacy of ADC189 tablets in the treatment of adult influenza subjects and determine the optimal therapeutic dose by analyzing the time of virus titer turning to negative. All the results will be used to design the Phase III study.
* Phase III study is to evaluate the efficacy of ADC189 tablets by analyzing the duration of remission of all influenza symptoms in adolescents and adults subjects with influenza.

Participants will be taken ADC189 teblets/Placebo once, and be observed by 22 days.

Phase II study has 3 groups: 15 mg ADC189; 45 mg ADC189; and Placebo; Phase III study has 2 groups: 45 mg ADC189; and Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years (including the cut-off point, Phase II) or 12 to 65 years (including the cut-off point, Phase III) with a body weight ≥ 20 kg, both sex;
2. Patients were diagnosed with Influenza A Virus Infection/Influenza B Virus Infection according to the following criteria: nasopharyngeal swab or oropharyngeal swab was positive under influenza rapid antigen test (RAT) (rapid influenza virus nucleic acid test or other rapid molecular diagnostic methods are also acceptable); and fever (ear temperature ≥ 37.3°C or axillary temperature ≥ 37.2°C), if taking antipyretics, ear temperature ≥ 37.3°C or axillary temperature ≥ 37.2°C after 4 hours taking antipyretics; at least one of the following symptoms are moderate or above (influenza symptom severity score ≥ 2) related to influenza: systemic symptoms: headache, fever or chills, muscle or joint aches, fatigue; respiratory symptoms: cough, sore throat, nasal congestion;
3. The time interval from the onset time of influenza to screening start ≤ 48 hours. Definition of influenza onset: the fever (ear temperature ≥37.3°C or axillary temperature ≥37.2°C or oral temperature ≥37.7°C) (ear temperature, axillary temperature and oral temperature measurements are acceptable), or the onset of any systemic symptoms or respiratory symptoms related to influenza;
4. Fertile subjects (including their partners) agree to take effective contraceptive methods throughout the study period and 3 months after study.
5. Voluntary participation in this clinical study and signing of the informed consent.

Exclusion Criteria:

1. Patients with known allergies to the test preparation, any of its components or related preparations (or severe allergic constitution), and who are judged by the investigator to have a safety risk for enter the trial;
2. Patients diagnosed as severe/critical flu at screening, as defined below:

   1. Severe cases are defined as those meeting one of the following conditions:

      High fever over 3 days, accompanied by severe cough, expectoration, bloody sputum, or chest pain; rapid breathing, dyspnea, and cyanosis of the lips; mental changes such as slow response, drowsiness, restlessness, or convulsions; severe vomiting, diarrhea, and dehydration; complicated with pneumonia; significant exacerbation of the original underlying disease;
   2. Critical cases are defined as those meeting one of the following conditions:

   Respiratory failure; acute necrotizing encephalopathy; shock; multiple organ dysfunction;
3. High-risk population in severe cases are defined as those meeting any of the following conditions, and who are judged by the investigator to have a safety risk in the trial:

   Patients with severe or poorly controlled underlying diseases, such as chronic respiratory diseases, liver diseases, chronic kidney diseases, severe hematological diseases, chronic congestive heart failure [New York Heart Association (NYHA) cardiac function classification III-IV], nervous system and neuromuscular diseases, metabolic diseases, etc.; Subjects with clinically significant abnormalities in the corrected QT interval (QTc> 450ms for males or QTc> 470ms for females) on electrocardiogram (QTcF calculated according to the Fridericia formula); Subjects with immunodeficiency, such as malignant tumor, organ or bone marrow transplantation, HIV infection, or taking immunosuppressants in the past 3 months; Subjects with other diseases requiring treatment with aspirin or salicylate drugs; Subjects with obesity [body mass index (BMI) greater than 30 kg/m2].
4. Subjects with a known history of dysphagia or any gastrointestinal disease that affects drug absorption (including but not limited to reflux esophagitis, chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, post-subtotal gastrectomy, etc.);
5. Subjects who had used anti-influenza virus drugs (oseltamivir, zanamivir, peramivir, favipiravir, arbidol, baloxavir, amantadine or rimantadine, etc.) within 2 weeks before screening or had received influenza vaccine within 6 months before screening;
6. Subjects with acute respiratory tract infection, otitis media, sinusitis or other infectious diseases such as bronchitis, pneumonia, tuberculosis or other infectious diseases within 2 weeks before screening;
7. Subjects with other bacterial or viral infections at the time of screening and need systemic antibacterial or antiviral treatment, or subjects with blood routine test: white blood cell count (WBC) > 10.0×109/L at the time of screening;
8. Pregnant or lactating women or positive pregnancy test. Pregnancy test is not required for women who have stopped menstruation for more than 2 years, confirmed postmenopausal women or women who have undergone hysterectomy, bilateral oophorectomy or tubal ligation surgery;
9. Suspected or confirmed history of alcohol or drug abuse;
10. Those who have participated in other drug clinical trials within 3 months before taking the drug;
11. Those who are not suitable for participation in the study in the judgment of the investigator.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
the severity of influenza | 22 days
  All subjects recorded 7 symptoms associated with influenza (cough, sore throat, headache, nasal congestion, fever or chills, muscle or joint pain, and fatigue) on a 4-point scale (0 points, none; 1 point, mild; 2 points, moderate; 3 points, severe) in a self-assessment on Dairy Card.
the safety of study drug | 22 days
  Collect all the Adverse Events during the whole study.

CONTACTS AND LOCATIONS:
Locations (1):
- Rui Jin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao J, Sheng G, Lyu Y, Sun Y, Wang S, Chen X, Ye F, Chen L, Xu X, Wang H, Wu B, Peng C, Deng M, Qu L, Jiang X, Hu J, Feng Y, Li Y, Peng J, Li W, Shao L, Gao F, Tian D, Tan J, Zheng H, Chen M, Wu H, Zhu X, Zhou M, Qu J. Oral ADC189 for adults and adolescents with uncomplicated influenza. J Infect. 2025 Apr;90(4):106472. doi: 10.1016/j.jinf.2025.106472. Epub 2025 Mar 13. PMID 40089214